CLINICAL TRIAL: NCT02096276
Title: Boostrix Pregnancy Registry: a Prospective, Exploratory, Cohort Study to Detect and Describe Any Abnormal Pregnancy Outcomes in Women Intentionally or Unintentionally Vaccinated With Boostrix® During Pregnancy or Within 28 Days Preceding Conception
Brief Title: Boostrix® Pregnancy Registry
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 201327
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Results first posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-11

CONDITIONS: Pertussis
Keywords: Pregnancy Registry; Boostrix; Women; Cohort; Prospective; Pregnancy outcome; Exploratory
MeSH Terms: conditions — Whooping Cough | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Exposure Group_Prospective: Pregnant women within the United States (US) who are exposed to Boostrix vaccine during pregnancy or within 28 days preceding conception and with known pregnancy outcomes. Reporting of exposed pregnancies is voluntary and prospective (i.e., registration to registry is done before the outcome of the pregnancy is known)
  Interventions: Other: Data collection
- Exposure Group_Retrospective: Pregnant women within the United States (US) who are exposed to Boostrix vaccine during pregnancy or within 28 days preceding conception and with known pregnancy outcomes. Reporting of exposed pregnancies is voluntary and retrospective (i.e., pregnancy outcome is already known at the time of registration to Registry)
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Initial and follow-up data will be collected using questionnaires.

SUMMARY:
The purpose of this Registry is to detect and describe any abnormal pregnancy outcomes, including teratogenicity, in females intentionally or unintentionally exposed to Boostrix during their pregnancies in the US. The Registry requires voluntary, prospective reporting of eligible pregnancies by patients and health care providers (HCPs). Data such as vaccination with Boostrix during pregnancy or within 28 days preceding conception, potential confounding factors (such as exposure to other medications) and information related to the outcome of the pregnancy will be collected prospectively

DETAILED DESCRIPTION:
The Registry was originally initiated on 03 May 2005, as part of a program of enhanced pharmacovigilance. Following new European Union Pharmacovigilance legislation, pregnancy registries are to be considered as post-authorization safety studies (PASS). The ongoing Registry will therefore be converted into a PASS study in Q1 2014.

Exposed pregnancies reported to the Registry before the transition into a PASS (between 03 May 2005 and Q1 2014), from which data were collected and analyzed prospectively, will also be included in the analyses.

Some pregnancy exposures may be reported after pregnancy outcome has been identified (retrospective reports). The Registry will capture retrospective reports, but these reports will not be included in the analyses of prospective reports.

Pregnancy outcome data will be collected using questionnaires within 2 months of the estimated date of delivery (EDD) and approximately 6 months and 12 months after the EDD (for all live births for whom the contact details of their HCP will be available) to ascertain the presence of birth defects not diagnosed before, from Q1 2014 to Q3 2019.

ELIGIBILITY:
Inclusion Criteria:

A subject will be included in the Registry if all of the following criteria are met:

* Exposure to vaccine occurs during pregnancy or within 28 days preceding conception.
* Subject is a US resident.
* A HCP is identified (name, address and phone number).
* Subject can be identified (by GSK or HCP).

Data from registered subjects will be included in the analyses if the following criterion is met:

• Pregnancy is ongoing and the outcome is unknown.

Exclusion Criteria:

Data from registered subjects will not be included in the analyses if the following criterion is met:

• Outcome of pregnancy is known at the time of initial report. Types of known outcomes include prenatal testing reports in which the results are abnormal or outside the reference range, indicating possible abnormality in the fetus. Typically, pregnancies > 16 weeks gestation will have undergone prenatal testing that can identify whether a child has congenital abnormalities.

Ages: 12 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Eligible pregnancies reported by patients and HCPs
Sampling Method: Non-Probability Sample
Enrollment: 1517 (Actual)
Dates: Start 2014-03-31 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total of 1517 pregnancy reports (1455 prospective and 62 retrospective) were collected in the Boostrix US Pregnancy Registry. Of the 1455 prospective reports, 250 had known pregnancy outcomes, 1188 were lost to follow-up and 17 pregnancies were ongoing. Of the 62 retrospective reports, 55 had known pregnancy outcomes and 7 were lost to follow-up.
Groups:
- Exposure Group_Prospective: Pregnant women within the United States (US) who were exposed to Boostrix vaccine during pregnancy or within 28 days preceding conception and with known pregnancy outcomes. Reporting of exposed pregnancies was voluntary and prospective (i.e., registration to registry was done before the outcome of the pregnancy is known)
- Exposure Group_Retrospective: Pregnant women within the United States (US) who were exposed to Boostrix vaccine during pregnancy or within 28 days preceding conception and with known pregnancy outcomes. Reporting of exposed pregnancies was voluntary and retrospective (i.e., pregnancy outcome was already known at the time of registration to Registry)
Period: Overall Study
Arm/Group | Exposure Group_Prospective | Exposure Group_Retrospective
Started | 250 | 55
Completed | 250 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exposure Group_Prospective | Exposure Group_Retrospective | Total
Number analyzed (Participants) | 250 | 55 | 305
Age, Customized [Count of Participants; unit: Participants] — Age Range is 13 - 42 Years for prospective cases and 14 - 40 Years for retrospective cases
  Participants
    Pregnant women (13-42 Years) | 248 | 28 | 276
    Unknown | 2 | 27 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 250 | 55 | 305
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Known Pregnancy Outcomes, by Type of Pregnancy Outcomes in Women Intentionally or Unintentionally Vaccinated With Boostrix During Pregnancy or Within 28 Days Preceding Conception.
Description: Pregnancy outcomes included live births, spontaneous abortions (pregnancy loss <22 weeks of gestation), stillbirths (pregnancy loss ≥22 weeks of gestation) and elective terminations.
  Each pregnancy outcome was further classified according to the presence or absence of a birth defect.
Time Frame: Data collected between 03 May 2005 to 02 August 2019: For each subject from date of registration until the pregnancy outcome documentation date (Exposure_Prospective group) or at pregnancy outcome documentation date (Exposure_Retrospective group)
Population: The analysis was performed on total cohort which included participants with known pregnancy outcomes.
Measure: Count of Participants; unit: Participants
Arm/Group | Exposure Group_Prospective | Exposure Group_Retrospective
Number analyzed (Participants) | 250 | 55
Participants
  Live birth without birth defects | 244 | 33
  Live birth with birth defects | 3 | 16
  Spontaneous abortion without birth defects | 3 | 1
  Spontaneous abortion with birth defects | 0 | 0
  Stillbirth without birth defects | 0 | 4
  Stillbirth with birth defects | 0 | 1
  Elective termination without birth defects | 0 | 0
  Elective termination with birth defects | 0 | 0

ADVERSE EVENTS:
Time Frame: Data collected between 03 May 2005 to 02 August 2019: For each subject from date of registration until the pregnancy outcome documentation date (Exposure_Prospective group) or at pregnancy outcome documentation date (Exposure_Retrospective group)
Description: Classification of events as SAE or other AE were unidentified. Pregnancy case reports were analyzed by case in scope of the Registry. Those cases may have had AEs co-reported. The systematic analysis of these AEs was not among the objectives of the study.
Arm/Group | Exposure Group_Prospective | Exposure Group_Retrospective
All-Cause Mortality (participants affected / at risk) | 3/250 | 6/55
Serious Adverse Events (participants affected / at risk) | 3/250 | 1/55
Other Adverse Events (participants affected / at risk) | 0/250 | 0/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exposure Group_Prospective (N=250) | Exposure Group_Retrospective (N=55)
Spontaneous abortion without birth defects (Pregnancy, puerperium and perinatal conditions) | 3 | 1 — Classification of this event as SAE or other AE was unidentified
Spontaneous abortion with birth defects (Pregnancy, puerperium and perinatal conditions) | 0 | 0 — Classification of this event as SAE or other AE was unidentified
Elective termination without birth defects (Pregnancy, puerperium and perinatal conditions) | 0 | 0 — Classification of this event as SAE or other AE was unidentified
Elective termination with birth defects (Pregnancy, puerperium and perinatal conditions) | 0 | 0 — Classification of this event as SAE or other AE was unidentified

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT02096276/Prot_SAP_000.pdf